CLINICAL TRIAL: NCT04465890
Title: Phase IIa Single Dose and Phase IIb Mutiple Dose Clinical Studies to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Subcutaneously Injected PD-L1 Antibody ASC22 in Patients With Chronic Hepatitis B
Brief Title: A Phase II Study of Subcutaneously Injected PD-L1 Antibody ASC22 in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other); Beijing Clinical Service Center (Other)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC-ASC22-II-CTP-01
Record Dates: First submitted 2020-06-22; First posted 2020-07-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-09

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis b (CHB); PD-L1; Fc fusion protein injection
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- cohort1: Single dose ASC22 injection 0.3mg/kg (Experimental): Single dose ASC22 Injection; Specification: 200mg/1ml/1bottle; Subcutaneous injection; once administration,0.3mg/kg dose of the drug once.
  Interventions: Drug: ASC22
- cohort2:Single dose ASC22 injection 1.0mg/kg (Experimental): Single dose ASC22 Injection; Specification: 200mg/1ml/1bottle; Subcutaneous injection; once administration,1.0mg/kg dose of the drug once.
  Interventions: Drug: ASC22
- cohort3:Single dose ASC22 injection 2.5mg/kg (Experimental): Single dose ASC22 Injection; Specification: 200mg/1ml/1bottle; Subcutaneous injection; once administration,2.5mg/kg dose of the drug once.
  Interventions: Drug: ASC22
- cohort4: Multiple dose ASC22 injection 1.0mg/kg (Experimental): Multiple dose ASC22 injection; Specification: 200mg/1ml/1bottle; Subcutaneously administered once every 2 weeks , 4 received 1.0mg/kg, up to 24 weeks
  Interventions: Drug: ASC22
- cohort5: Multiple dose ASC22 injection 2.5mg/kg (Experimental): Multiple dose ASC22 injection; Specification: 200mg/1ml/1bottle; Subcutaneously administered once every 2 weeks , 4 received 2.5mg/kg, up to 24 weeks
  Interventions: Drug: ASC22
- cohort4: Placebo sodium chloride injection A (Placebo Comparator): Placebo saline injection; Specification: 90mg/10ml/1 bottle; Subcutaneously administered every 2 weeks (Q2W, known as one drug administration cycle), duration: once every 2 weeks (Q2W), up to 12 weeks. Based on the weight of the patients, an equal dose of placebo was administered according to the incoming dose group (1.0mg/kg).
  Interventions: Drug: sodium chloride
- cohort5: Placebo sodium chloride injection B (Placebo Comparator): Placebo saline injection; Specification: 90mg/10ml/1 bottle; Subcutaneously administered every 2 weeks (Q2W, known as one drug administration cycle), duration: once every 2 weeks (Q2W), up to 12 weeks. Based on the weight of the patients, an equal dose of placebo was administered according to the incoming dose group (2.5mg/kg).
  Interventions: Drug: sodium chloride
- cohort6: Multiple dose ASC22 injection 1.0mg/kg (Experimental): Multiple dose ASC22 injection; Specification: 200mg/1ml/1bottle; Subcutaneously administered once every 2 weeks , 4 received 1.0mg/kg, up to 24 weeks
  Interventions: Drug: ASC22
- cohort6: Placebo sodium chloride injection A (Placebo Comparator): Placebo saline injection; Specification: 90mg/10ml/1 bottle; Subcutaneously administered every 2 weeks (Q2W, known as one drug administration cycle), duration: once every 2 weeks (Q2W), up to 12 weeks. Based on the weight of the patients, an equal dose of placebo was administered according to the incoming dose group (1.0mg/kg).
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: ASC22 — 200mg/1ml/1bottle
  Arms: cohort1: Single dose ASC22 injection 0.3mg/kg; cohort2:Single dose ASC22 injection 1.0mg/kg; cohort3:Single dose ASC22 injection 2.5mg/kg; cohort4: Multiple dose ASC22 injection 1.0mg/kg; cohort5: Multiple dose ASC22 injection 2.5mg/kg; cohort6: Multiple dose ASC22 injection 1.0mg/kg
Drug: sodium chloride — 90mg/10ml/1 bottle
  Arms: cohort4: Placebo sodium chloride injection A; cohort5: Placebo sodium chloride injection B; cohort6: Placebo sodium chloride injection A

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ASC22 in the treatment of chronic hepatitis B after single and multiple drug administration.

DETAILED DESCRIPTION:
The study consists of two parts: the ASC22 single-dose IIa study and the ASC22 multi-dose IIb study. The IIa study consists of 3 cohorts of 0.3mg/kg, 1.0mg/kg and 2.5mg/kg, and the IIb study consists of 2 cohorts of 1.0mg/kg and 2.5mg/kg. The objective is to evaluate the safety, tolerance and efficacy of ASC22 in patients with chronic hepatitis B (CHB), and to provide a guidance for the determination of dosage regimen.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old (including boundary value), gender unlimited；
2. Chronic hepatitis B patients with clear diagnosis of Hematology, etiology and clinical (for example: HBsAg positive for more than 6 months);
3. HBV-DNA turns negative after treatment with nucleoside (acid) drugs;
4. cohort1-5:HBsAg≤ 10000 IU/mL; cohort6: HBsAg≤ 100 IU/mL;
5. HBeAg negative;
6. The fertile female subjects or the fertile male subjects agreed to take contraceptive measures from 7 days before the first administration until 24 weeks after the end of the administration cycle of ASC22. The serum pregnancy test of fertile female subjects must be negative within 7 days before the first administration.

Exclusion Criteria:

1. Patients with hepatitis a, hepatitis c (HCV RNA>15IU/L), hepatitis d or HIV infection; Patients with other active infections (e.g., respiratory tract infection, urinary tract infection and herpes simplex, cytomegalovirus, epstein-barr virus);
2. Fibrosis stage: Cirrhosis, portal hypertension, or advanced fibrosis (defined as Fibroscan≥9.5kPa or ARFI≥1.81m/sec or Fibrosis-4 (FIB-4)≥3.25 or METAVIR F≥3);
3. Liver cancer patients or blood AFP>1×ULN;
4. cohort1-5：Patients who received interferon therapy within 6 months before the first administration; cohort6: Patients who received interferon therapy before the first administration;
5. Patients receiving immunosuppressive therapy within 3 months before the first administration (except interferon);
6. The investigator judges that the participants are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the decreased HBsAg levels at 12 or 24 weeks of treatment or at 4, 12, or 24 weeks of follow-up visits compared with baseline. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).
Evaluate the number of patients with ≥0.5log reduction in HBsAg log10IU/ mL at 12 or 24 weeks of treatment, or at 4, 12, or 24 weeks of follow-up visits compared with baseline. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).

SECONDARY OUTCOMES:
Evaluate the decline value of HBsAg level. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).
Evaluate the propotion's change of HBsAg < 0.05IU/ml in each cohort. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).
Evaluate the changes of cytokines (IL-2, IFN-γ) in each cohort. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).
Evaluate the changes of peripheral blood lymphocyte subsets in each cohort. | 48 weeks
  Each multiple dose cohort will last 48 weeks (24-weeks treatment plus 24-weeks follow up).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided